CLINICAL TRIAL: NCT04421638
Title: Drug Hypersensitivity Reactions To Cephalosporins
Brief Title: Cephalosporin Hypersensitivity
Acronym: CephALL
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0021
Record Dates: First submitted 2020-01-08; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-04

CONDITIONS: Drug Hypersensitivity
Keywords: Drug Hypersensitivity Reaction; Drug Provocation Test; Cephalosporins; Betalactams; Risk Factor
MeSH Terms: conditions — Drug Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background :

Although the hypersensitivity reactions to cephalosporins have been recently a more focused subject, studies on the cephalosporin as an allergen are significantly less frequent that those regarding penicillins. Most of the available data regards cephalosporin sensitization in patients previously allergic to penicillin. Like penicillins, cephalosporins represent one of the most prescribed classes of antibiotics. The diagnosis of cephalosporin hypersensitivity is based mainly on clinical history, skin tests (ST) and drug provocation tests (DPT). This succession of tests, performed in specialized services, allows to eliminate responsibility for the drug in many cases (80-85%). The drug allergy work-up also allows to identify profiles of allergy to cephalosporins, with different patterns of cross-reactivity.

Objective: To analyse the characteristics of patients studied in our Unit for suspicion of cephalosporin hypersensitivity.

Methods: This retrospective study will comprise all the patients who attended the allergy service of the UH of Montpellier from 1997 till 2018 with a clinical history evocative of cephalosporin drug hypersensitivity reaction (DHR), who underwent a drug allergy work up and who gave their consent to be included in the study . The Patients are selected from the Drug Allergy & Hypersensitivity Database (DAHD).

ELIGIBILITY:
Inclusion criteria:

- Patients with one or more ST and DPT tests to cephalosporins

Exclusion criteria:

- Patients refusing to take part in the study

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient consulting in our allergy unit for a suspicion of DHR to cephalosporins and who underwent a drug allergy work-up.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Identify clinical variables associated with allergy to cephalosporins | 1 day
  Identify clinical variables associated with allergy to cephalosporins

SECONDARY OUTCOMES:
Determine the risk variables associated with allergy to cephalosporins | 1 day
  Determine the risk variables associated with allergy to cephalosporins
To calculate the negative predictive value of cephalosporin DTP | 1 years
  In the subgroup of patients for whom we have data on readministration of a negatively tested cephalosporin following drug allergy work-up, we will calculate the negative predictive value of cephalosporin DPT.

CONTACTS AND LOCATIONS:
Overall Officials: Anca Chiriac, MD,PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided